CLINICAL TRIAL: NCT03663153
Title: SEMA4C as a Relapse Biomarker in Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: Hubei Cancer Hospital (Other); Qilu Hospital of Shandong University (Other); Wuhan Central Hospital (Other); Xiangyang Central Hospital (Other); The First People's Hospital of Jingzhou (Other); The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Clinical Professor, Tongji Hospital
Other Study IDs: 2018-TJ-BCP
Record Dates: First submitted 2018-09-03; First posted 2018-09-10 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SEMA4C high value follow-up group: Postoperative SEMA4C value is higher than 5.00 ng/ml.
  Interventions: Other: SEMA4C high value follow-up group
- SEMA4C low value follow-up group: Postoperative SEMA4C value is lower than 5.00 ng/ml.
  Interventions: Other: SEMA4C low value follow-up group

INTERVENTIONS:
Other: SEMA4C high value follow-up group — Serum samples will be collected every 3 months for the first year after surgery and then every 6 months to first progression defined as death or recurrence of the breast cancer or until 5 years since last patient in, whichever occurs first. Imaging examination and biopsy or surgery if necessary are recommended for patients with elevated SEMA4C. Serum SEMA4C levels will be tested in single center in order to decrease bias and be measured using a double antibody sandwich ELISA method using in-house SEMA4C detection kits.
  Groups: SEMA4C high value follow-up group
Other: SEMA4C low value follow-up group — Serum samples will be collected every 3 months for the first year after surgery and then every 6 months to first progression defined as death or recurrence of the breast cancer or until 5 years since last patient in, whichever occurs first. Imaging examination and biopsy or surgery if necessary are recommended for patients with elevated SEMA4C. Serum SEMA4C levels will be tested in single center in order to decrease bias and be measured using a double antibody sandwich ELISA method using in-house SEMA4C detection kits.
  Groups: SEMA4C low value follow-up group

SUMMARY:
Breast cancer remains the most common cancer in women worldwide. Semaphorin4C (SEMA4C) has previously been identified as a highly expressed protein by breast cancer-associated lymphatic endothelial cells (LECs). The objective of this study is to investigate SEMA4C's potential role as an early relapse biomarker in breast cancer.

DETAILED DESCRIPTION:
Breast cancer remains the most common cancer in women worldwide, with approximately 1.68 million new cases, and 0.52 million deaths, annually. Meanwhile the incidence of breast cancer continues to increase. Although regular clinical examination, mammography, ultrasonography, and magnetic resonance imaging can detect some recurrence patients, the lack of robust biomarkers for monitoring of anti-tumor therapies and detection of recurrence reduce the treatment effectiveness of current strategies for breast cancer.

Semaphorin4C (SEMA4C) has been previously identified as a highly expressed protein by breast cancer-associated lymphatic endothelial cells (LECs) using in situ laser capture microdissection of lymphatic vessels, followed by cDNA microarray analysis. Moreover, membrane-bound SEMA4C is cleaved by matrix metalloproteinase (MMPs) to release a soluble form of this protein. The study is undertaken to explore SEMA4C's potential role as an early relapse biomarker in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed new diagnosis of breast cancer according to biopsy or surgery

Exclusion Criteria:

* Patients who are not mentally capable of giving written informed consent
* Serum samples doesn't qualified
* Patients who refuse follow-up on their conditions
* Patients with prior cancer history
* Patients with a diagnosis of other severe acute or chronic medical may increase the risk associated with study participation or may interfere with the interpretation of the study results and, in the judgement of the Investigator, would make the patient inappropriate for enrollment in this study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants including patients with breast cancer. All cases were confirmed histopathologically according to the WHO Classification of Tumors.
Sampling Method: Non-Probability Sample
Enrollment: 4200 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy (sensitivity, specificity, positive predictive value, negative predictive value) of SEMA4C in predicting recurrence of breast cancer | 5 years
  Analyze the sensitivity, specificity, positive predictive value, negative predictive value, accuracy of SEMA4C in predicting recurrence of breast cancer

SECONDARY OUTCOMES:
Disease Free Survival | 5 years
  Disease Free Survival (DFS) can be determined according to clinical practice based on any of the following: applicable imaging technique, biopsy and surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Qinglei Gao, MD, PhD, Principal Investigator — Tongji Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wei JC, Yang J, Liu D, Wu MF, Qiao L, Wang JN, Ma QF, Zeng Z, Ye SM, Guo ES, Jiang XF, You LY, Chen Y, Zhou L, Huang XY, Zhu T, Meng L, Zhou JF, Feng ZH, Ma D, Gao QL. Tumor-associated Lymphatic Endothelial Cells Promote Lymphatic Metastasis By Highly Expressing and Secreting SEMA4C. Clin Cancer Res. 2017 Jan 1;23(1):214-224. doi: 10.1158/1078-0432.CCR-16-0741. Epub 2016 Jul 8. PMID 27401250
- [Background] Gurrapu S, Pupo E, Franzolin G, Lanzetti L, Tamagnone L. Sema4C/PlexinB2 signaling controls breast cancer cell growth, hormonal dependence and tumorigenic potential. Cell Death Differ. 2018 Jul;25(7):1259-1275. doi: 10.1038/s41418-018-0097-4. Epub 2018 Mar 19. PMID 29555978